CLINICAL TRIAL: NCT05749770
Title: Hormonal Contributors to Coronavirus SARS-CoV-2 Infection (COV-ENDO)
Brief Title: Hormonal Contributors to COVID-19 Infection (COV-ENDO)
Acronym: COV-ENDO
Status: Completed | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 05C021
Record Dates: First submitted 2023-02-20; First posted 2023-03-01 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: COVID-19 Pandemic; Endocrine System Diseases
MeSH Terms: conditions — COVID-19; Endocrine System Diseases | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, whole blood and DNA samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- COVID-19: Patients affected with SARs-CoV-2 infection and hospitalized in the COVID wards of Auxologico
  Interventions: Other: blood testing
- CONTROLS: 440 NON-COVID subjects collected retrospectively at other collaborating centers) University of Siena, Campus Biomedico Rome, University of Catania, San Giovanni Rotondo)
  Interventions: Other: blood testing

INTERVENTIONS:
Other: blood testing — blood testing for basal hormones and markers of inflammation
  Other Names: thyroid US scan in case of thyroid dysfunctions

SUMMARY:
The goal of this observational study is to measure the changes in the parameters of endocrine function and tissue sensitivity to hormones induced by SARs-CoV-2 infection.

The main questions it aims to answer are:

* Does SARs-CoV-2 infection causes endocrine dysfunctions?
* Does the treatment of the underlying endocrine dysfunctions, improves the clinical outcome or the occurrence of late onset complications of SARs-CoV-2 infection?
* Are patients with previously known endocrine diseases more fragile in case of SARs-CoV-2 infection? Participants will undergo blood testing and a physical examination at admission, during hospitalization at discharge and 3 and 6 moths after discharge They results will be compared to those of patients admitted for other reasons in order to assess whether the prevalence of endocrine dysfunctions is increased compared with controls.

DETAILED DESCRIPTION:
The objectives of the study are the following:

Primary objectives:

1. to measure endocrine function tests in patients affected by COVID-19, in order to evaluate whether SARs-CoV-2 causes endocrine alterations and whether endocrine diseases/dysfunctions correlate with the severity of SARs-CoV-2 infection and mortality.
2. to evaluate whether genetic variants in the sex-steroid or vitamin D (VDR) nuclear receptors or ACE are more prevalent in patients with SARs-CoV-2 infection than controls.
3. to evaluate whether vitamin D supplementation in subjects with vitamin D deficiency may influence the outcome of SARs-CoV-2 infection
4. To correlate the influence of overweight/obesity/neck circumference with the evolution of SARs-CoV-2 infection

Secondary objectives:

Correlate the endocrine function tests with patients' age, disease's outcome, markers of inflammation.

The identification of endocrine conditions associated with a worse outcome of SARs-CoV-2 infection, would identify significant risk factors to be reduced/prevented in these patients. For example, if endocrine patients will result more fragile in case of infection, we could systematically screen some parameters and early treat associated defects in order improve the outcome of SARs-CoV-2 infection.

ELIGIBILITY:
Inclusion Criteria:

* Nasal swab positive for Sars-CoV-2
* Moderate to severe respiratory dysfunction due to COVID-19, requiring hospitalization.

Exclusion Criteria:

* History of thyroid diseases before admission
* History of adrenal diseases
* History of hypogonadism (primary/secondary)
* History of pituitary diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a pilot study aiming at evaluating all the subjects with COVID-19 admitted to the Istituto Auxologico during pandemic.
  It is expected to recruit at least 220 COVID-19 subjects and 440 controls subjects collected retrospectively at the other centers.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Endocrine function and markers of inflammation: TSH | through study completion, an average of 1 year
  Change in TSH (thyroid stimulating hormone), mU/L
Endocrine function and markers of inflammation: IL-6 | through study completion, an average of 1 year
  Change in IL-6 (interleukin-6), U/L
Endocrine function and markers of inflammation: Testosterone | through study completion, an average of 1 year
  Change in total and free calculated testosterone, nmol/l
Endocrine function and markers of inflammation: Cortisol | through study completion, an average of 1 year
  Change in cortisol, ug/dl
Endocrine function and markers of inflammation: Reactive C-protein | through study completion, an average of 1 year
  Change in reactive C protein, mg/dl
Endocrine function and markers of inflammation: ACTH | through study completion, an average of 1 year
  Change in ACTH (Adrenocorticotropic hormone), pg/ml
Endocrine function and markers of inflammation: 25-OH vitamin D | through study completion, an average of 1 year
  Change in 25-OH vitamin D, ng/ml
Prevalence of genetic variants of target genes | through study completion, an average of 1 year
  NGS/direct sequence of androgen receptor (AR), progesterone receptor (PGR), estrogen receptors (ESR1 and 2), vitamin D receptor (VDR), Angiotensin-converting enzyme 2 (ACE2)
Effect of vitamin D deficiency | through study completion, an average of 1 year
  Assessment of the following parameters of clinical outcome: mortality, complication during hospitalization, complication after discharge, quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Luca Persani, MD, PhD, Principal Investigator — Istituto Auxologico Italiano IRCCS
Locations (1):
- Istituto Auxologico Italiano IRCCS, Milan, Italy

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in this topic. Data or samples shared will be coded, with no protected health information included. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis
Access Criteria: Access to individual participant data (IPD) can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).
URL: https://zenodo.org/records/5882276

REFERENCES:
- [Background] Campi I, Gennari L, Merlotti D, Mingiano C, Frosali A, Giovanelli L, Torlasco C, Pengo MF, Heilbron F, Soranna D, Zambon A, Di Stefano M, Aresta C, Bonomi M, Cangiano B, Favero V, Fatti L, Perego GB, Chiodini I, Parati G, Persani L. Vitamin D and COVID-19 severity and related mortality: a prospective study in Italy. BMC Infect Dis. 2021 Jun 14;21(1):566. doi: 10.1186/s12879-021-06281-7. PMID 34126960
- [Background] Campi I, Bulgarelli I, Dubini A, Perego GB, Tortorici E, Torlasco C, Torresani E, Rocco L, Persani L, Fugazzola L. The spectrum of thyroid function tests during hospitalization for SARS COV-2 infection. Eur J Endocrinol. 2021 May;184(5):699-709. doi: 10.1530/EJE-20-1391. PMID 33683214
- Available data/document: Individual Participant Data Set — https://zenodo.org/records/5913009